CLINICAL TRIAL: NCT05418712
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled Study Evaluating the Effects of VX-150 on C-Nociceptor Action Potentials in Healthy Subjects
Brief Title: A Microneurography (MNG) Study of VX-150 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VX22-150-012
Record Dates: First submitted 2022-06-09; First posted 2022-06-14 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Participants will receive placebo matched to VX-150.
  Interventions: Drug: Placebo
- VX-150 (Experimental): Participants will be randomized to receive a single dose of one of different dose levels VX-150.
  Interventions: Drug: VX-150

INTERVENTIONS:
Drug: Placebo — Placebo matched to VX-150 for oral administration.
  Arms: Placebo
Drug: VX-150 — Solution or Suspension for oral administration.
  Arms: VX-150

SUMMARY:
The purpose of this study is to determine if C fiber conduction is impacted by NAV1.8 modulation.

DETAILED DESCRIPTION:
This clinical trial information was submitted voluntarily under the applicable law and, therefore, certain submission deadlines may not apply. (That is, clinical trial information for this applicable clinical trial was submitted under section 402(j)(4)(A) of the Public Health Service Act and 42 CFR 11.60 and is not subject to the deadlines established by sections 402(j)(2) and (3) of the Public Health Service Act or 42 CFR 11.24 and 11.44.).

ELIGIBILITY:
Key Inclusion Criteria:

* Body mass index (BMI) of 18.0 to 30.0 kilogram per meter square (kg/m^2)
* A total body weight >50 kg

Key Exclusion Criteria:

* Participants who have any 1 of the following criteria in the foot/ankle in which MNG will be performed:

  * Injection of local anesthetics or steroids within 35 days prior to randomization
  * Unsuitable anatomy of the superficial peroneal nerve (i.e., nerve cannot be seen or palpated at the dorsum of the foot/ankle)
  * Infection, disease (dermatologic or vascular), ongoing pain, or recent trauma or surgery that may affect study assessments
* History of febrile illness within 14 days before study drug dosing
* Any condition possibly affecting drug absorption
* Participants with Type 1 or Type 2 diabetes mellitus
* Any dermatological (generalized) or autoimmune disease that may affect C-nociceptor excitability

Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2022-06-16 (Actual); Primary Completion 2022-09-14 (Actual); Study Completion 2022-09-23 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in Action Potential (AP) Latency at 0.25 Hertz (Hz) Over Time | From Baseline up to 3 Hours After Dose

SECONDARY OUTCOMES:
Change From Baseline in Percentage Slowing Over Time | From Baseline up to 3 Hours After Dose
  Percentage slowing is measured by a relative change in latency from the start to the end of each activity-dependent slowing (ADS) stimulus train.
Change From Baseline in the Time to Reverse 50 Percent (%) of the Activity-induced Latency Change After the End of Each ADS Stimulus Train Over Time | From Baseline up to 3 Hours After Dose
Change From Baseline in the Percentage Recovery of the Activity-induced Latency Change at 30 Seconds After the End of Each ADS Stimulus Train Over Time | From Baseline up to 3 Hours After Dose
Change From Baseline in Conduction Velocity at 0.25 Hz Over Time | From Baseline up to 3 Hours After Dose
Change From Baseline in AP Amplitude at 0.25 Hz Over Time | From Baseline up to 3 Hours After Dose
Change From Baseline in the Area Under the AP Peaks at 0.25 Hz Over Time | From Baseline up to 3 Hours After Dose
Safety and Tolerability as Assessed by Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAE) | Day 1 up to Day 10

CONTACTS AND LOCATIONS:
Locations (1):
- MAC Clinical Research, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/independent-research/clinical-trial-data-sharing